CLINICAL TRIAL: NCT00174057
Title: The Role of TSH Receptor, PPAR-r, IGF-1R, IGF and Cytokines in Different Stages of Graves'Ophthalmopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700644
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Graves' Ophthalmopathy
Keywords: Graves' ophthalmopathy; real time PCR; cytokines; Tsh receptor
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The exact mechanism of the pathogenesis of Graves' ophthalmopathy is still unknown. Histopathologically, extraocular muscle inflammation and orbital fat inflammation are two prominent changes. In the past year, we had investigated the morphological features of the Müller muscle in patients with thyroid lid retraction using the special stain and immunohistochemistry. In our findings, the smooth muscle cells, in the diseased group, were replaced by variable adipose and fibrosis tissues.

In recent years, TSHR, has been verified to express in orbital connective tissue and extra-ocular muscle. From functional studies and an increase in adipogenesis in cultured fibroblasts with expression of TSHR protein, the role not only the target but effector cells in orbital fibroblasts were validated. Quantitative RT-PCR may help to differentiate whether a less extent of expression at the end stage or low protein amount to be detected.

In recent years, the diverse phenotypes of orbital fibroblasts, with regard to expression of Thy-1 protein or not, had been reported from several studies, the investigators believed heterogeneity in orbital fibroblast may determine the clinical presentation of Graves'ophthalmopathy. We also are curious to know if the phenotypic heterogeneity of the fibroblasts in the ocular adnexal and orbital tissues correlates to distinct morphological features of adipogenesis and fibrosis.

Moreover, increased CD40 expression in skin fibroblasts were noted from patients with systemic sclerosis. Expression of IGF-I and IGF-IR seemed to be up-regulated in processes of several fibrotic diseases. A nuclear transcription factor, PPAR-γ, has been verified to have a close relationship with adipogenesis. We hypothesize that some immunological processes involve the ocular adnexal and orbital tissues, which result in various ophthalmological manifestations.

The purpose of this study is to investigate the different stage of the ocular adnexal and orbital tissues to identify the pathogenesis of Graves' ophthalmopathy by frozen sections with Immunohistochemistry, mRNA expression of TSH receptor, PPAR-γ, IGF-1R, and IGF-1 and different cytokines using quantitative RT-PCR and flow cytometry at the acute and stable stage in GO.

DETAILED DESCRIPTION:
The exact mechanism of the pathogenesis of Graves' ophthalmopathy (GO) is still unknown. Histopathologically, extraocular muscle inflammation due to lymphoid infiltration, edema and interstitial fibrosis, and increased glycosaminoglycan deposition and orbital fat inflammation are two prominent changes. There are various manifestations including ocular adnexal tissues inflammation, proptosis, lid retraction, extraocular movement limitation and compressive optic neuropathy. In the past year, we had investigated the morphological features of the Müller muscle in patients with thyroid lid retraction using the special stain and immunohistochemistry in formalin-fixed paraffin-embbeded (FFPE) sections. In our findings, the smooth muscle cells, in the diseased group, were replaced by variable adipose and fibrosis tissues. Two distinct features in the disease group seem to be notable for further investigation.

In recent years, TSHR, a putative autoantigen, has been verified to express in orbital connective tissue and extra-ocular muscle. In addition, they were further demonstrated to express on the surface of cultured orbital fibroblasts and orbital adipose tissue, in patients with GO in several laboratories. From functional studies and an increase in adipogenesis in cultured fibroblasts with expression of TSHR protein, the role not only the target but effector cells in orbital fibroblasts were validated7. We used immunohistochemistry to verify the existence of TSHR on the fibroblasts within the Müller muscle, and the positive staining is manifested in only18 % of patients. It may due to a less extent of expression at the end stage. We are very curious to know if there any difference on the expression of TSHR between orbital specimens from patients with acute and those with stable stage. Quantitative RT-PCR may help to differentiate whether a less extent of expression at the end stage or low protein amount to be detected.

In recent years, the diverse phenotypes of orbital fibroblasts, with regard to expression of Thy-1 protein or not, had been reported from several studies, the investigators believed heterogeneity in orbital fibroblast may determine the clinical presentation of Graves' ophthalmopathy. We also are curious to know if the phenotypic heterogeneity of the fibroblasts in the ocular adnexal and orbital tissues correlates to distinct morphological features of adipogenesis and fibrosis. In addition, systemic or local pro-inflammatory cytokines may contribute to turn on and turn off the expression of different roles of the fibroblasts.

Moreover, increased CD40 expression in skin fibroblasts were noted from patients with systemic sclerosis. Expression of IGF-I and IGF-IR seemed to be up-regulated in processes of several fibrotic diseases. A nuclear transcription factor, PPAR-γ, has been verified to have a close relationship with adipogenesis. In our previous study, the smooth muscle cells, in the diseased Mullers' muscle, were replaced by variable adipose and fibrosis tissues. The increased adipose and fibrosis tissue ex vivo of the Müller' muscle may result from over-action of some biochemical markers in the fibroblasts infiltrating around muscle cells. We hypothesize that some immunological processes involve the ocular adnexal and orbital tissues, which result in various ophthalmological manifestations.

The purpose of this study is to investigate the different stage ( acute or stable stage) of the ocular adnexal and orbital tissues ( including orbital fat, extraocular muscles, orbicularis muscles and eyelid fat) to identify and validate the pathogenesis of Graves ophthalmopathy by frozen sections of the ocular adnexal and orbital tissues with Immunohistochemistry (IHA) (Thy-1 and PPARγ), mRNA expression of TSH receptor, PPAR-γ, IGF-1R, and IGF-1 and different cytokines (IL-1β, IL-4, IL-6, IL-8) using quantitative RT-PCR and flow cytometry at the acute and stable stage in GO.

ELIGIBILITY:
Inclusion Criteria:patients with Graves ophthalmopathy -

Exclusion Criteria:no

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Shu Lang Liao, MD, Study Director — National Taiwan University Hospital
Locations (1):
- Shu Lang Liao, Taipei, Taiwan